CLINICAL TRIAL: NCT06177002
Title: SARS-CoV-2, TESTOSTERONE AND MALE FRAGILITY (PROTEGGIMI): A MULTIDIMENSIONAL RESEARCH PROJECT
Brief Title: SARS-CoV-2, TESTOSTERONE AND MALE FRAGILITY
Acronym: PROTEGGIMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Andrea Salonia, Prof, IRCCS San Raffaele
Other Study IDs: PROTEGGIMI - 01/2020
Record Dates: First submitted 2023-12-18; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: COVID-19; Testosterone Deficiency; Infertility, Male
MeSH Terms: conditions — COVID-19; Infertility, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Male COVID-19 patients: Male patients with an age > 18 affected by COVID-19 with biological samples positive for SARS-CoV-2 but with negative test
  Interventions: Diagnostic Test: Collection of biological data
- male healthy individuals: Healthy donors with an age> 18 accessing the IRCCS OSR Blood Donor Center
  Interventions: Diagnostic Test: Collection of biological data

INTERVENTIONS:
Diagnostic Test: Collection of biological data — Biological sample will be collected from the COVID19 patients and from healthy donors

SUMMARY:
The hormonal environment (steroid, primarily) could have a very relevant pathophysiological role in association with SARS-CoV-2. That is, testosterone could play a relevant role in leaving male subjects more exposed to infection and more prone to developing severe complications following COVID-19 infection.

DETAILED DESCRIPTION:
Preliminary data suggests that male individuals are more susceptible to COVID-19 infection, at least in Western countries, and that their mortality rate is higher than female individuals. This would seem to suggest that the hormonal environment (steroid, primarily) could have a very relevant pathophysiological role in association with SARS-CoV-2. That is, testosterone could play a relevant role in leaving male subjects more exposed to infection and more prone to developing severe complications following COVID-19 infection. Another option is that COVID-19 infection could cause a condition of acute hypogonadism, following which, the exhaustion of androgenic action could act as a co-trigger of a severe or even fatal course of the disease.

ELIGIBILITY:
Inclusion Criteria:

Patient Cohort:

* Male patients with an age > 18 hospitalized in the departments dedicated to the care of patients affected by COVID-19 at the San Raffaele Hospital and with:
* biological samples positive for SARS-CoV-2;
* negative test but highly suggestive clinical and radiological picture;
* patients discharged from the emergency room with biological samples positive for SARS-CoV-2;
* ability to read and sign the informed consent

Control Cohort:

* healthy donors with an age> 18 accessing the IRCCS OSR Blood Donor Center;
* ability to read and sign the informed consent

Exclusion Criteria:

* People with an age < 18;
* incapacity to read and sign the informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Males
Study Population: Male COVID-19 patients and male healthy individuals
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-05-19 (Actual); Primary Completion 2025-05-18 (Estimated); Study Completion 2025-05-18 (Estimated)

PRIMARY OUTCOMES:
Dosage of the androgenic hormonal environment in the blood of patients and healthy controls | Baseline

SECONDARY OUTCOMES:
create an international (European) registry for the management of sensitive data in epidemiological terms and pathology outcomes relating to males with confirmed COVID-19 infection and age-matched healthy controls | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No